CLINICAL TRIAL: NCT01291446
Title: Objective Markers Flatulence: Determination of Gas Production and Evacuation in Response to Dietary Manipulations
Brief Title: Effect of Diet on Intestinal Gas Production and Evacuation in Healthy Subjects and Flatulent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PR(AG)32/2010
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Flatulence
Keywords: Intestinal gas production; Intestinal microbiota
MeSH Terms: conditions — Flatulence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High flatulogenic diet (Sham Comparator): 3-day diet containing fermentable residues
  Interventions: Dietary Supplement: High flatulogenic diet

INTERVENTIONS:
Dietary Supplement: High flatulogenic diet — During 3-days subjects will consume a diet with high content of fermentable residues

SUMMARY:
Background Some patients complain of excessive evacuation, which may become socially disabling (Azpiroz F & Malagelada J-R, 2005). However, there no systematic investigation on the range of gas evacuation in healthy subjects and in subjects complaining of flatulence under basal conditions and in response to a high-flatulogenic diet (Azpiroz F & Levitt DG, 2009).

Hypothesis Patients complaining of excessive passage of gas per anus have more intestinal gas production and more anal gas evacuation during basal conditions and in response to a high flatulogenic diet than healthy subjects. This abnormality is related to the differences in colonic microflora.

Objectives

* To determine the normal range of intestinal gas evacuation under basal conditions and in response to a high flatulogenic diet.
* In patients complaining of flatulence, to determine whether intestinal gas evacuation under basal conditions and in response to a high flatulogenic diet is increased.
* To identify differences in the microbiota pattern in subjects with normal and excessive anal gas evacuation.
* In patients complaining of flatulence, to determine the segmental distribution of intestinal gas after a diet challenge.

Methods Healthy subjects (n=20) and patients complaining of flatulence (n=30) will undergo a 3-day basal phase on their current diet and a 3-day challenge phase on a high-flatulogenic diet; patients will be followed-up for 7 days on a low-flatulogenic diet. The following g measurements will be performed: daily measurement of the number of anal gas passages with an event marker, continuous recording of anal gas evacuation in the laboratory using an electronic leakage-free gas collection system, colonic flora analysis by fecal sampling, and segmental gas distribution in the gut by abdominal computer tomography (CT) imaging.

Relevance These studies will allow to develop the normal range of anal gas evacuation during basal conditions. Furthermore, a provocative test will be developed for the diagnosis of excessive gas production in patients complaining of flatulence. This data will allow a proper diagnosis of these patients and will pave the path for a rational management and for the development of evidence-based treatment strategies. This pilot study will allow a proper design with adequate sample size calculation in future interventional studies.

DETAILED DESCRIPTION:
Background Some patients complain of excessive evacuation, which may become socially disabling (Azpiroz F & Malagelada J-R, 2005). However, the physiology and pathophysiology of flatulence remains poorly understood (Azpiroz F & Levitt DG, 2009).

Gas evacuated by anus originates by-and-large in the colon, where unabsorbed meal residues are fermented by colonic bacteria (Anderson et al., 1981;Levitt et al., 1987;Flourie et al., 1988). Indeed, it has been shown that some food components are incompletely absorbed in the small bowel and enter the colon (Wolever & Robb, 1992;Grimble, 1989;Steggerda FR, 1968;Wagner et al., 1977;Steggerda F.R. & Dimmick, 1966;Stone-Dorshow & Levitt, 1987;Wursch et al., 1989) and that other intraluminal substrates interfere with the absorption of nutrients (Boibin M et al., 1998;Hamberg et al., 1989;Brugge & Rosenfeld, 1987;Taylor et al., 1986;Layer et al., 1986). Hence, the volume of gas production and anal evacuation is determined by two main factors: the diet, particularly the amount of fermentable residues, and the individual composition of colonic microflora. Within subjects, gas output varies in relation to the diet (Steggerda FR, 1968;Kirk, 1949). However, there is a great interindividual variability, and gas evacuation in subjects maintained on a similar diet may differ substantially.

It has been shown that healthy subjects on a normal diet containing 200 g of beans evacuate 705 mL gas per 24 hours, whereas with a fiber the diet gas evacuation was 214 mL (Tomlin et al., 1991). In healthy subjects the frequency of gas evacuation is variable, usually around 10 evacuation per day (Furne & Levitt, 1996). Based on observations on a patient that who passed large amounts of flatus, a classification of foodstuffs depending on their gas producing capacity was elaborated (Sutalf LO & Levitt MD, 1979). Few studies on specific foodstuffs have been later added to complement this information (Wolever & Robb, 1992;Wagner et al., 1977;Hickey C et al., 1972). However, there no systematic investigation on the range of gas evacuation in healthy subjects and in subjects complaining of flatulence under basal conditions and in response to a high-flatulogenic diet.

Procedures Recruitment questionnaire A questionnaire will be used to evaluate gas evacuation, bowel habit and functional gut symptoms.

Daily measurement of the number of anal gas evacuations and symptoms The number of gas evacuations per anus will be measured using an event marker during daytime. At the end of the day the following parameters will be recorded on a questionnaire: discomfort related to flatulence and evaluation of abdominal discomfort/pain (using 0-10 analogue scales); the number of bowel movements and form (using the Bristol scale; (Heaton & O'Donnell, 1994) and gastrointestinal well-being (satisfaction/dissatisfaction using a 10 point scale graded from +5 to -5).

Analysis of colonic flora The composition of the intestinal flora will be evaluated measuring flora composition in stools. Subjects will be supplied with two Stool Collecting Kits (each containing two weighed sampling tubes containing RNA synthesis stabilization buffers (RNA later, Ambion), one of which is a spare) into which they will provide a small sample of their stool (at least 30g). After mixing the stool with the buffer in the supplied tube, subjects will store the tubes in the box at home until they next visit at the hospital, where it will be centrifuged at 12000rpm for 5 minutes, supernatant removed and fecal pellet stored at - 80oC in the Gastroenterology Research Unit. Samples will be transported to Danone Research, France where they will be analysed for composition of intestinal flora (bacteria).

Using molecular based methods, the concentration of dominant and some sub-dominant bacterial groups of intestinal flora will be measured. These include bacteria that belong to Actinobacteria, Bacteroidetes, Firmicutes, Fusobacteria, Proteobacteria, Euryarcheota groups.

Continuous recording of anal gas evacuation Participants will be studied in the laboratory. After a standard breakfast, rectal gas will be collected via a rectal cannula. Anal gas will be collected via a leak proof, low resistance collection line, using a barostat and the volume will be continuously recorded for either 3 or 8 hours (see study design). The composition of the gas collected will be analyzed.

Once the subjects are positioned in bed, a non-stretch belt, 48 mm wide, with a metric scale will be adjusted around the abdomen by means of two elastic bands. All girth changes will be measured while the subjects are breathing relaxed, and will be referenced to the mid point of respiratory displacements.

A graded questionnaire will be used to measure the intensity and the type of sensations perceived, and an anatomical questionnaire to measure the location and extension of the perceived sensations. The graded questionnaire includes five visual analogue scales graded from 0 (no perception) to 6 (pain), specifically for scoring: a) sensation of increased abdominal pressure, b) sensation of abdominal distension, c) colicky/rumbling sensation, d) puncture/stinging sensation, and d) other type of sensation (to be specified by the participant in the questionnaire), respectively. The questionnaire includes two additional scales for scoring feeling of difficult evacuation of gas per anus, and belching, respectively, that will be analyzed separately. Subjects will be asked to score any perceived sensation (one or more perceived simultaneously) on the scales. The anatomical questionnaire incorporates a diagram of the abdomen divided in nine regions corresponding to epigastrium, periumbilical area, hypogastrium, both hypochondria, flanks, and ileal fossae. Subjects will be instructed to mark the location, i.e., abdominal region (s) or extraabdominal, where the sensations are perceived.

Segmental gas distribution in the gut In patients complaining of bloating, an abdominal CT scan will be taken. This scan will be used to rule out organic disorders. Furthermore, using an original program, abdominal morpho-volumetric analysis will be performed to measure gas volumes in different gut. All female participants with childbearing potential will undergo a urine pregnancy test 24 hours prior to the scan.

Hyperflatulogenic diet challenge For 3 days participants will be asked to consume a diet rich in fermentable residues to increase their gas production rate.

Low-flatulogenic diet At the end of the study, patients will be put on a low residue diet for 7 days; this will give an indication of the potentially expected response to treatment.

Working Plan Each subject will attend the following visits; the first recruitment visit will be performed by the attending physician in the outpatient clinic, and the rest, including the physiological measurements in the Digestive System Research Unit; CT imaging will be performed in the Department of Radiology.

Visit 1. Recruitment: entry questionnaires. Visit 2. Before basal period: instructions, informed consent, and delivery of event marker, questionnaires, and material for fecal sampling.

Visit 3. Last day of basal phase. Continuous recording of anal gas evacuation. Delivery of dietary instructions (high-flatulogenic diet) and questionnaires. In 8 patients segmental gas distribution will be also measured during the basal phase.

Visit 4. Last day of challenge phase. Continuous recording of anal gas evacuation. CT for evaluation of segmental gas distribution in the gut. In patients only: delivery of dietary instructions (low-flatulogenic diet) and questionnaires.

Visit 5. Last day of correction phase. In patients only: collection of data and materials.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between the ages of 18 and 70 years.
* Excessive gas evacuation will be checked at the first visit with a questionnaire "do you pass too much gas per anus, i.e., a lot of a passages along the day ?"
* Subjects of normal body weight or with overweight ie not obese (body mass index between 18 and 30 kg/m2, bounds included )
* Subject willing to maintain their current diet without significant changes (ie. new caloric restriction or elimination diet) for the duration of the study
* Subjects who provide written informed consent before participating in the study after being given a full description of the study

Exclusion Criteria:

* Subjects with abnormal finding of vital signs at the screening examination which would interfere with the objectives of the study
* Subjects with a history of clinical significant hepatic, renal, respiratory, psychiatric, neurological, endocrine, infectious, cardiovascular, pulmonary, haematological or systemic disorders.
* Antecedents of abdominal surgery, excluding appendicectomy or hernia
* Subjects who are already taking or have taken in the past 2 months any investigational drug
* Use of antibiotics in the month preceding the inclusion visit.
* Current use of any medications with potential central nervous system effects as judged by the investigator (including but not limited to antidepressants, anxiolytics, opiate pain medications)
* Taking drugs that might modify gastrointestinal function
* Taking antibiotics within 60 days prior to entry into the study.
* Subjects with a history of drug, alcohol or other substance abuse (including caffeine and tobacco), or other factors limiting their ability to co-operate during the study.
* Subjects not willing or not available to attend all the test-days and investigations as foreseen by the protocol.
* Subjects not collaborating, unable to understand the aim, the procedure or the possible hazards of the study.
* Patient with allergy or hypersensitivity to food proposed during the food challenge

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Intestinal gas evacuation | 7 days
  Intestinal gas evacuation will be measured during a 3-day basal phase on their current diet and a 3-day challenge phase on a high flatulogenic diet

SECONDARY OUTCOMES:
Colonic microbiota pattern | 7 days
  Colonic microbiota pattern will be measured during a 3-day basal phase on their current diet and a 3-day challenge phase on a high flatulogenic diet

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital, Barcelona 08035, Spain
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain